CLINICAL TRIAL: NCT03642964
Title: A Phase 2a Study to Evaluate the Safety, Tolerability and Initial Efficacy of Pramipexole IR, Given With Ondansetron in Patients With Major Depressive Disorder
Brief Title: A Study in Patients With Major Depressive Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTC-003
Record Dates: First submitted 2018-07-05; First posted 2018-08-22 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): CTC-501 (pramipexole IR, given with ondansetron) given orally twice daily
  Interventions: Drug: CTC-501
- placebo (Placebo Comparator): generic placebo tablets given orally twice daily
  Interventions: Drug: CTC-501

INTERVENTIONS:
Drug: CTC-501 — pramipexole IR, given with ondansetron

SUMMARY:
This is a Phase 2a, placebo-controlled, single-blind study in up to 24 patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
This is a Phase 2a, placebo-controlled, single-blind study in up to 24 patients with major depressive disorder (MDD).

Subjects will sign consent form prior to any study related procedure and will complete screening assessments. Subjects will be randomized to either the treatment group or the placebo group at a ratio of 1:1.

The study will be conducted in two parts. Titration period On Day 1, subjects will complete all baseline assessments prior to the 1st dosing.

Pramipexole group: Consenting individuals meeting accession criteria will start pramipexole 2.0mg daily dose (1.0mg twice a day) with ondansetron 16mg daily dose (8mg twice a day). Pramipexole will be titrated up daily or every two days depends on each patients' tolerability up to the first intolerable dose (FID) or maximum allowed dose (5 mg/day) according to titration schedule (Table 1). Once subjects reach their FID, their maximum allowed dose (MTD) will be defined as 1 mg below their FID.

During titration, subjects will be admitted to the clinic (subjects will be discharged on the day following their pramipexole FID or Day 8 if subjects reach to 5 mg/day of pramipexole.

Placebo group will take 3 placebo tablets twice a day. Maintenance period During the maintenance phase, patients will be treated with pramipexole MTD or MAD with ondansetron 16mg/day for the remainder of the 8-week treatment.

Placebo group is taking 3 tablets of placebo twice a day during the trial. Exit visit After the Week 8 visit, study medications will be discontinued, and subject will return for Exit visit at Week 9.

After the Exit visit, all subjects will return to their prior treatment for depression or started on a new therapeutic regimen as medically appropriate.

At study completion (or at other times in accordance with Stopping Rules given below), and all study participants will return to their pre-admission therapeutic regimen or started on a new therapeutic regimen as medically appropriate. Higher doses of pramipexole IR may be tapered off at rates deemed medically appropriate by PI.

In this modified single blind study, efficacy raters will be kept unaware of the participants' treatment status.

An independent data and safety monitoring board (DSMB) will be appointed to have responsibility for safeguarding the interests of the trial subjects and assessing the safety and tolerability of the study treatments during the trial.

ELIGIBILITY:
Inclusion Criteria:

- Patient Population: Males and females with a diagnosis of major depressive disorder

Inclusion Criteria:

1. Signed an Institutional Review Board (IRB) approved informed consent document indicating that they understand the purpose of and procedures required by the study and are willing to participate in the study and comply with all study procedures and restrictions. Informed consent must be obtained from the patient and/or a designated representative prior to initiating screening procedures to evaluate eligibility of the study.
2. Males and females aged 18 and 65 years inclusive.
3. Meet DSM-V R criteria for major depression, single episode or recurrent episode, with or without melancholia and without psychotic features (296.21, 296.22, 296.23, 296.31, 296.32, or 296.33).
4. Had a total score of > 18 on the HAM-D (17-item version), and a score of > 2 on the depressed mood item of the HAM-D at the screening visit and at the baseline visit.
5. Patients who are currently not on any antidepressants or, Patients on antidepressants and agree to the appropriate washout period (certain antidepressants with prolonged effects (e.g., fluoxetine) may need longer than 2 weeks post-discontinuation to obtain relatively uncontaminated baseline evaluation).
6. Agreed not to start psychotherapy or behavior therapy during the trial. Patients currently on these types of therapy for at least 3 months are eligible for the study and could continue to receive therapy during the trial.

Exclusion Criteria:

1. Women who are pregnant, or lactating; or taking a low-estrogen "mini-pill" contraceptive.
2. Individuals who are currently taking either study medication (pramipexole and/or ondansetron).
3. Renal and hepatic dysfunction with:

   * Total Bilirubin: >1.5 x UNL
   * AST: >2.5 x UNL
   * ALT: >2.5 x UNL
   * Serum Creatinine: >1.5 x UNL
   * Creatinine Clearance: <30 mL/min (calculated by Cockcroft and Gault equation)
4. Hypersensitivity to any component of either study medication.
5. Lifetime history of hypomania/mania, psychotic disorder, dementia and borderline or antisocial personality disorders.
6. History of a serious suicidal attempt in the past 12 months; presence of serious suicidal tendencies/potential; modified C-SSRS >4.
7. Positive urine screen for benzodiazepines, cocaine/cocaine metabolites, cannabinoids, amphetamines, barbiturates, and opiates or history of moderate or severe substance dependence (drugs or alcohol, DSM-V-R criteria) within the past 6 months of the screening visit.
8. Non-responders to at least two trials of antidepressant treatment in the past. (Therapeutic dose for at least 6 weeks)
9. Patients currently taking or have taken the following medications within the past 6 months.

   * Centrally acting dopamine antagonists
   * MAOI
10. Patients considered unlikely to co-operate in the study, and/or poor compliance anticipated by the investigator.
11. Patients who have clinical significant hypotension or any clinical significant ECG abnormality at screening.
12. Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.
13. Patients who have participated in another clinical trial with an investigational drug within previous 30 days or 5 half-lives whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability will be assessed by the determination of a Maximum Tolerated Dose of pramipexole | multiple over 8 weeks
  All subjects will be assessed for dose limiting side effects such as nausea, vomiting and diarrhea.

SECONDARY OUTCOMES:
Safety will be assessed by Incidence of Treatment-Emergent Adverse Events | Multiple over 8 weeks
  Incidence and nature of adverse events; vital signs; weight ; physical examination changes; clinical laboratory evaluations; ECG.
The Montgomery-Åsberg Depression Rating Scale | Multiple over 7 weeks
  Change from baseline in the following depression scale; The Montgomery-Åsberg Depression Rating Scale (abbreviated MADRS) is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorder. Mean change from baseline on the Montgomery Asberg Depression Rating Scale. (MADRS) Relative to Standard of Care. The MADRS is a 10 item scale with each item scored from 0 to 6 where 0 represents minimal symptoms and 6 represents maximum response to that item. The total MADRS score ranges from 0 to 60.
Clinical Global Impression - Severity scale | Multiple over 7 weeks
  Change from baseline in the following depression scales.Mean change from baseline on the CGI-Severity of Illness(CGI-SI) score overtime.The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  o CGI-Global Improvement (CGI-GI) score at the end of 8-week maintenance period
Clinical Global Impression - Improvement scale | at week 8 only
  Change from baseline in the following depression scales;The Clinical Global Improvement - CGI-Global Improvement (CGI-GI) score at the end of 8-week maintenance period is a one question scale comparing who the clinician feels the patient's condition has changed from baseline. The scale is from 0-7 (0 being 'not assessed' to 7 being 'very much worse'.
Pharmacokinetics will measure plasma concentrations of pramipexole and ondansetron | Multiple over 7 weeks
  Plasma concentrations of pramipexole and ondansetron will be measured at various times throughout the study in only pramipexole group. Both groups will have blood draws.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Leibowitz, MD, Principal Investigator — Collaborative Neuroscience Network
Locations (1):
- Collaborative Neuroscience Network, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share IPD.